CLINICAL TRIAL: NCT01637077
Title: RC11C3, Pilot Placebo-controlled Evaluation of Pregabalin as a Means to Prevent the Paclitaxel-Associated Acute Pain Syndrome
Brief Title: Pregabalin in Preventing Acute Pain Syndrome in Patients Receiving Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC11C3; NCI-2011-03646 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT02166385 (obsolete NCT alias)
Record Dates: First submitted 2012-03-09; First posted 2012-07-10 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Pain; Peripheral Neuropathy
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (pain therapy) (Experimental): Patients receive pregabalin PO BID, beginning on the first night of chemotherapy, for 12 weeks and then QD for 1 week.
  Interventions: Drug: pregabalin; Other: questionnaire administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID, beginning on the first night of chemotherapy, for 12 weeks and then QD for 1 week.
  Interventions: Drug: placebo; Other: questionnaire administration

INTERVENTIONS:
Drug: pregabalin — Given PO
  Other Names: 3-Isobutyl GABA; CI-1008; Lyrica; PD-144723
  Arms: Arm I (pain therapy)
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies pregabalin in preventing acute pain syndrome in patients receiving paclitaxel. Pregabalin may control the pain caused by cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To obtain pilot data regarding the possible effect of pregabalin on pain related to paclitaxel-associated acute pain syndrome (P-APS). SECONDARY OBJECTIVES: I. To obtain pilot data regarding the possible effect of pregabalin on paclitaxel-induced peripheral neuropathy. II. To obtain pilot data regarding the possible relative toxicities related to pregabalin therapy in this study situation. TERTIARY OBJECTIVES: I. To characterize neurological testing abnormalities that might occur with the P-APS, and to evaluate neurological testing abnormalities during the period of the longer-term chemotherapy-induced peripheral neuropathy (CIPN). II. To determine the PRO incidence and characteristics of, and change in, P-APS and paclitaxel induced more chronic CIPN over several cycles. These data will serve to confirm the results obtained in our previous natural history study N08C1. OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive pregabalin orally (PO) twice daily (BID), beginning on the first night of chemotherapy, for 12 weeks and then once daily (QD) for 1 week. ARM II: Patients receive placebo PO BID, beginning on the first night of chemotherapy, for 12 weeks and then QD for 1 week. After completion of study treatment, patients are followed up every 30 days for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* Ability to complete questionnaires by themselves or with assistance Paclitaxel at a dose of 80 mg/m^2 given, in the adjuvant setting, every week for a planned course of 12 weeks without any other concurrent therapy
* Paclitaxel at a dose of 80 mg/m2 given, in the adjuvant (postoperative or neo-adjuvant) setting, every week for a planned course of 12 weeks without any other concurrent cytotoxic chemotherapy (trastuzumab and/or other antibody and/or small molecule treatment is allowed, except for PARP inhibitors).
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Negative pregnancy test (serum or urine) done =< 7 days prior to registration, for women of childbearing potential only (per clinician discretion)

Exclusion Criteria:

* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception since this study involves agents that have known genotoxic, mutagenic and teratogenic effects
* Previous diagnosis of diabetic or other peripheral neuropathy
* Current, planned or previous use, within last 6 months, of gabapentin or pregabalin
* History of allergic or other adverse reactions to gabapentin or pregabalin
* Significant renal insufficiency with a history of a creatinine clearance (CrCL) < 30ml/min
* Prior exposure to neurotoxic chemotherapy
* Seizure history
* Diagnosis of fibromyalgia
* Previous exposure to paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Cancer Center of Kansas, Wichita, Kansas
  - Essentia Health-Duluth CCOP, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Pregabalin): Patients receive pregabalin (75 mg (one capsule)) PO BID, beginning on the first night of chemotherapy, for 12 weeks and then QD for 1 week.
- Arm II (Placebo): Patients receive placebo (one capsule) PO BID, beginning on the first night of chemotherapy, for 12 weeks and then QD for 1 week.
Period: Overall Study
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Started | 23 | 23
Completed | 19 | 22
Not Completed | 4 | 1
Not completed — Cancel | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No cycle 1 questionnaire data | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (12.9) | 53.2 (14.3) | 53.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Worst of the Pain Scores for the Week Following the First Cycle of Paclitaxel Administration, Paclitaxel-associated Acute Pain Syndrome (P-APS) Pain Score
Description: Worst of the pain scores for the week following the first cycle of paclitaxel administration, as measured by a question on the daily post-paclitaxel questionnaire. Worst pain over the first 6 days following treatment initiation. Higher scores represent more pain (0: No aches or pains -10: Aches or pains as bad as can be).
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
units on a scale | 2.6 (2.5) | 3.2 (3.0)
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.56, Kruskal-Wallis

2. Primary Outcome: Maximum of the Average Pain Scores (Item 3, Appendix IV) Over the Period From Treatment Initiation to Day 7 (for Cycle 1).
Description: Maximum of average pain scores over 6 days following initiation of treatment. Average pain over the first 6 days following treatment initiation. Maximum of the average pain scores (item 3, appendix IV; "Please rate the same aches/pain by circling the ONE number that best describes your aches/pains on the AVERAGE in the last 24 hours.") over the period from treatment initiation to day 7 (for cycle 1). Higher scores represent more pain (0: No aches or pains -10: Aches or pains as bad as can be).
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
units on a scale | 2.6 (2.2) | 2.2 (2.6)
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.48, Kruskal-Wallis

3. Secondary Outcome: Area Under the Curve Per Assessment (aAUCpa) of Worst, Average and Least Pain (Items 1-3 Appendix IV) for the First Cycle of Treatment.
Description: Average Area Under the Curve per assessment (aAUCpa) of worst, average, and least pain (items 1-3 app. IV; "Please rate any aches/pains that are NEW since your last dose of paclitaxel, and that you think might be related to your chemotherapy treatment by circling ONE number that best describes your aches/pains at its WORST in the last 24 hours.", "Please rate the same aches/pains by circling the ONE number that best describes your aches/pains at its LEAST in the last 24 hours.", "Please rate the same aches/pain by circling the ONE number that best describes your aches/pains on the AVERAGE in the last 24 hours.") for the first cycle of treatment. Scores are reported on a 0-100 scale, where 100=better outcome QOL. The aAUCpa is the average of each AUC between each sequential assessment from treatment-initiation to the day-6 assessment.
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Population: The number analyzed for average pain over the past 24 hours differs from the overall number analyzed due to missing data.
Measure: Mean (Standard Deviation); unit: average(subscale value*assessment)
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
average(subscale value*assessment)
  Worst pain over the past 24 hours | 80.7 (22.3) | 82.6 (24.0)
  Average pain over the past 24 hours: number analyzed (Participants) | 18 | 22
  Average pain over the past 24 hours | 82.8 (20.2) | 86.8 (19.7)
  Least pain over the past 24 hours | 82.6 (23.0) | 91.3 (14.8)
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Worst pain over the past 24 hours; Test type: Superiority; p = 0.62, Kruskal-Wallis
Statistical Analysis 2: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Average pain over the past 24 hours; Test type: Superiority; p = 0.22, Kruskal-Wallis
Statistical Analysis 3: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Least pain over the past 24 hours; Test type: Superiority; p = 0.07, Kruskal-Wallis

4. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events Considered At Least Possibly Related to Treatment
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Baseline, day 8 prior to each paclitaxel course, and then every 30 days for 6 months after completion of study treatment
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 2.2 | 0

5. Secondary Outcome: The Percentage of Patients Who Use Non-prescription Pain Medications
Description: The percentage of patients who use non-prescription pain medications are reported by arm below.
Time Frame: From treatment initiation to 6 months.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 52.6 | 50
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.87, Chi-squared

6. Secondary Outcome: The Percentage of Patients Taking Opioid Medications
Description: The percentage of patients taking opioid medications are reported below by arm.
Time Frame: From treatment initiation to 6 months.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 15.8 | 18.2
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.84, Chi-squared

7. Secondary Outcome: The Percentage of Patients Who Report the Development of New Aches/Pains That They Attribute to Paclitaxel
Description: The percentage of patients who report the development of new aches/pains that they attribute to paclitaxel in the first week of chemotherapy are reported by arm below.
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 23.5 | 59.1
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.03, Chi-squared

8. Secondary Outcome: The Worst Pain Reported at the End of the Week for the Overall Week (Item 2 Appendix V)
Description: The worst pain reported at the end of the week for the overall week ("New aches and pains at their worst over the past week") are reported below. This question was only supposed to be answered by patients who responded "yes" to the first question. Currently, all responses are included, regardless of whether the patient should've responded or not. The worst pain reported at the end of the week for the overall week (item 2 appendix V: "Please rate any aches/pains that you have by circling ONE number that best describes your aches/pains at its worst over the last week.") Higher scores represent more pain (0: No aches or pains -10: Aches or pains as bad as can be).
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
units on a scale | 2.4 (2.1) | 4.7 (3.2)
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.12, Kruskal-Wallis

9. Secondary Outcome: The Percentage of Patients Who Report, at Week's End, Using Non-prescription Pain Medications
Description: The percentage of patients who report, at week's end, using non-prescription pain medications ("Have you used non-prescription meds like aspirin, Tylenol, Motrin, Ibuprofen, or Advil over the past week?") are reported by arm below. This question was only supposed to be answered by patients who responded "yes" to the first question. Currently, all responses are included, regardless of whether the patient should've responded or not.
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 66.7 | 60.
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.78, Chi-squared

10. Secondary Outcome: The Percentage of Patients Who Report, at Week's End, Using Opioids
Description: The percentage of patients who report, at week's end, using opioids ("Have you used opioids like codeine, oxycodone, or morphine for this pain over the past week?") are reported by arm below. This question was only supposed to be answered by patients who responded "yes" to the first question. Currently, all responses are included, regardless of whether the patient should've responded or not.
Time Frame: From treatment initiation to 6 days following treatment initiation; up to 7 days
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage of patients | 0 | 26.7
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Test type: Superiority; p = 0.16, Chi-squared

11. Secondary Outcome: Area Under the Curve (AUC) of EORTC Sensory, Autonomic, and Motor Neuropathy Subscales
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neurophathy Module (EORTC QLQ-CIPN20) Sensory, Autonomic, and Motor Neuropathy Subscales. The EORTC CIPN20 scoring algorithm was used for the sensory (items 31-36, 39, 40 and 48), motor (items 37, 38, 41-45, 49), and autonomic (items 46, 47, 50) subscale scores on a 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for each subscale is calculated as the average of each AUC between each sequential assessment from treatment-initiation to the 6-month assessment. For example; for each patient and each subscale, the subscale values at treatment-initiation and assessment-1 are used to calculate an Area Under the Curve (AUC) for that assessment time-period. Then these AUCs for all available assessment time-periods up to 6-months are averaged to yield the aAUCpa per patient per subcale.
Time Frame: From treatment initiation to 6 months.
Measure: Mean (Standard Deviation); unit: average(subscale value*assessment)
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
average(subscale value*assessment)
  Sensory | 88.4 (12.5) | 84.5 (16.7)
  Autonomic | 88.4 (17.6) | 88.6 (15.8)
  Motor | 92.0 (11.0) | 90.2 (10.7)
Statistical Analysis 1: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Sensory neuropathy; Test type: Superiority; p = 0.46, Kruskal-Wallis
Statistical Analysis 2: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Autonomic neuropathy; Test type: Superiority; p = 0.86, Kruskal-Wallis
Statistical Analysis 3: Comparison: Arm I (Pregabalin) vs Arm II (Placebo); Motor neuropathy; Test type: Superiority; p = 0.40, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Time Frame: Baseline, day 8 prior to each paclitaxel course, and then every 30 days for 6 months after completion of study treatment
Description: The revised NCI Common Terminology Criteria for AE (CTCAE) version 4.0 will be utilized for AE reporting. Cancels and Withdrawal by Subject in the Participant Flow table did not receive treatment. Serious AE (SAE) reports for this study may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited Adverse Events (EAEs), and appear in the SAE table.
Arm/Group | Arm I (Pregabalin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/22
Other Adverse Events (participants affected / at risk) | 15/21 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pregabalin) (N=21) | Arm II (Placebo) (N=22)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pregabalin) (N=21) | Arm II (Placebo) (N=22)
Hearing impaired (Ear and labyrinth disorders) | 2 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (54) | 14 (35)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 8 (34) | 13 (74)
Fatigue (General disorders) | 1 (2) | 2 (8)
Pain (General disorders) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (13) | 3 (15)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (10) | 3 (3)
Dizziness (Nervous system disorders) | 5 (27) | 6 (29)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No